CLINICAL TRIAL: NCT07149948
Title: Teen motHers' ReproductIve and behaVioral Health intErvention in Barbados (THRIVE)
Brief Title: Teen motHers' ReproductIve and behaVioral Health intErvention in Barbados
Acronym: THRIVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hada Fongha Ieong, PhD (Other)
Collaborators: Rotary Club of Barbados (Unknown)
Responsible Party: Sponsor-Investigator, Hada Fongha Ieong, PhD, Principal Investigator and Sponsor-Investigator, Ross University School of Medicine
Organization: Ross University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RUSM20240405-CANREC20250903
Record Dates: First submitted 2025-08-11; First posted 2025-09-02 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy in Adolescence
Keywords: Integrated care; Barbados; Caribbean health; Psychoeducation; Community-based intervention; Global Health; THRIVE; Adolescent Pregnancy; Teenage Mothers; Parenting; Reproductive Health; Mental Health; School Reentry; Family Planning Services; Contraceptive Use; Low-Income Population; Behavioral Health; Anxiety; Depression
MeSH Terms: conditions — Psychological Well-Being; Anxiety Disorders; Depression | interventions — Nicotine

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the THRIVE integrated care intervention group or the standard care control group, and each group will receive their respective care in parallel throughout the study period.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, care providers, and outcomes assessors will not be informed of group assignments. Randomization and assignment will be handled by third-party study personnel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THRIVE Integrated Care Intervention (Experimental): Participants in this arm will receive the THRIVE integrated reproductive and behavioral health intervention, consisting of seven biweekly psychoeducation modules delivered in-person or via Zoom. The program addresses reproductive health knowledge, parenting skills, mental health, substance use, and life skills to prevent repeat adolescent pregnancy.
  Interventions: Behavioral: THRIVE Integrated Care Program
- Standard Care Control (No Intervention): Participants in this arm will receive standard postnatal and psychosocial care provided by community health centers in Barbados, such as health check-ups and basic social support services. They will not receive the THRIVE modules.

INTERVENTIONS:
Behavioral: THRIVE Integrated Care Program — The THRIVE Integrated Care Program is a psychoeducational behavioral intervention for adolescent mothers that combines reproductive health education and mental health support. It includes seven biweekly in-person or virtual sessions covering topics such as sexual health, parenting, mental health, substance use prevention, social support, and professional development. The intervention is delivered by trained medical students and staff using interactive learning modules and assessments.
  Other Names: THRIVE
  Arms: THRIVE Integrated Care Intervention

SUMMARY:
The goal of this clinical trial is to learn if an integrated care program can help improve overall health and prevent repeat pregnancy in teen mothers in Barbados. The study focuses on young women ages 10 to 25 who became pregnant during their teenage years and are experiencing stress or mood-related symptoms. This study is currently pending ethics committee review and has not yet begun enrolling participants.

The main questions it aims to answer are:

* Does the THRIVE program improve participants' mental health and parenting skills?
* Does the program help prevent repeat, unplanned pregnancies?

Researchers will compare participants who receive the THRIVE program to those who receive standard care to see if the program leads to better physical and emotional health.

Participants will:

* Take part in seven biweekly in-person or virtual sessions focused on reproductive and behavioral health;
* Complete health checks and questionnaires about their mood, parenting stress, and support;
* Receive follow-up contact after the sessions are completed.

The THRIVE program includes education on sexual health, mental health, parenting, and life skills. Participants will receive small incentives and support throughout the study. All study activities will begin only after full ethics approval is obtained.

DETAILED DESCRIPTION:
Teen pregnancy remains a significant public health concern in many parts of the world, including Latin America and the Caribbean (LAC). Young mothers in these regions often experience high rates of repeat, unplanned pregnancies, mental health challenges, limited educational opportunities, and reduced access to reproductive and behavioral health care. Despite the need, there are few published, evidence-based interventions targeting this population in the Caribbean, and even fewer that take a holistic, integrated approach.

This study introduces THRIVE - Teen motHers' ReproductIve and behaVioral health intErvention - a novel, integrated care program designed to support the overall health and development of young mothers in Barbados who became pregnant during adolescence. The THRIVE program provides education and support in both reproductive and behavioral health, recognizing that these domains are deeply interconnected in the lives of young mothers.

The study is a randomized controlled trial (RCT). It is designed to assess whether the THRIVE intervention improves participants' mental health, parenting confidence, and reproductive health outcomes compared to standard care. It also aims to reduce the risk of repeat adolescent pregnancy and promote engagement in school or professional development.

Background and Rationale Studies in high-income countries have shown that teen pregnancy prevention efforts are most effective when they include empowerment through education and psycho-social support. However, in LAC regions such as Barbados, there is a lack of published evidence on whether similar approaches can be successfully adapted and implemented. Many existing programs narrowly focus on a single health domain (e.g., sexual health education or treatment of depressive symptoms) and often overlook the broader context of a teen mother's life, including parenting stress, family support, and barriers to education or employment.

THRIVE was developed in response to this gap. It is a culturally appropriate, multidimensional intervention that integrates reproductive and behavioral health education tailored specifically for young mothers in Barbados. This study seeks to generate scientific evidence on the feasibility, acceptability, and preliminary effectiveness of THRIVE, laying the foundation for future longitudinal studies in the region.

Study Design This is a two-arm, randomized controlled, double-blinded Phase 0 clinical trial involving a total of 50 participants, with 25 randomized to the THRIVE intervention group and 25 to the control group receiving standard care. Participants are young women between the ages of 10 and 25 who became pregnant between the ages of 10 and 19, are from low-income households (defined as an annual income of ≤ BDS $20,000 or USD ~$10,000), and report mood-related symptoms such as sadness or lack of interest following childbirth.

Intervention: THRIVE Program

The THRIVE intervention group will participate in seven biweekly sessions, delivered either in person at accessible community sites (e.g., Rotary Club of Barbados) or via virtual conferencing platforms. Each session includes:

* A brief health check (e.g., vital signs)
* A 40-minute interactive psychoeducation module
* A 15-minute assessment and feedback session

The THRIVE curriculum integrates topics across five key domains:

* Reproductive Health Education - contraception, safe sex, STI prevention
* Behavioral Health Support - managing stress, anxiety, depression, and mood
* Parenting Skills - building confidence in parenting, positive discipline
* Social Support - identifying and using family and community resources
* Professional Development - goal setting, school re-engagement, job readiness

Each module includes clear learning objectives, practical tools, and opportunities for self-reflection. Participants are encouraged to apply what they learn between sessions. They will also receive light snacks, printed materials, and regular follow-up contact.

The control group will continue receiving the usual care provided through local clinics or community partners. They will undergo the same assessments as the intervention group but will not receive any THRIVE modules.

Study Objectives and Outcomes The primary objective of the study is to evaluate whether the THRIVE intervention improves young mothers' overall health, mood, and parenting skills. The secondary objective is to assess whether the program reduces the likelihood of repeat, unintended pregnancy and improves participants' engagement with school or professional opportunities.

Researchers will assess outcomes through structured interviews and validated measurement tools at baseline and follow-up. The measures include:

* Mental health symptoms (depression, anxiety, stress)
* Parenting attitudes and behaviors
* Use of contraception and reproductive health practices
* Social support
* School or job engagement
* Repeat pregnancy incidence (as self-reported)

All participants will complete assessments via structured interviews administered by trained research assistants or volunteer medical students. The data will be collected using secure digital tools and analyzed using statistical methods appropriate for small randomized trials.

Participant Support and Ethical Considerations The THRIVE study has been designed to prioritize the dignity, safety, and autonomy of participants. Written informed consent will be obtained from all participants. For those under 18, both parental/guardian consent and participant assent will be required.

Participants are free to withdraw from the study at any time without consequence. The research team is trained to identify signs of distress, abuse, or unsafe situations, and will provide referrals to appropriate services if needed.

To support participation, all individuals who complete study assessments will receive an incentive. Snacks and drinks will also be provided during in-person sessions. Participants in both groups will be treated with equal respect and receive the same level of follow-up care and attention.

This study will be conducted in accordance with the latest version of the Declaration of Helsinki and is currently pending reviewing and approval by the Institutional Review Board (IRB) of Ross University School of Medicine. The THRIVE protocol also adheres to national and institutional ethical standards for research involving human participants.

Innovation and Community Impact THRIVE represents one of the first published, structured interventions of its kind in the Caribbean. It integrates health, education, and psychosocial care into one coordinated program - a unique model in this context. The study will not only address the immediate needs of participants but will also contribute data to help shape public health policy and practice in the Caribbean and beyond.

Through partnerships with local clinics, schools, and organizations such as the Rotary Club of Barbados, the THRIVE study strengthens community capacity for supporting vulnerable young mothers and promotes intergenerational health improvement.

The findings will be shared with local stakeholders and published in peer-reviewed journals to expand the body of knowledge on adolescent pregnancy prevention in low- and middle-income countries (LMICs).

Future Directions

While this is a pilot study, the long-term goal is to use findings from THRIVE to:

* Inform the development of larger-scale interventions and cohort studies
* Guide educational and health policy initiatives across the LAC region
* Establish best practices for integrated care models for adolescent mothers

The THRIVE model has the potential to be adapted to other LAC countries and similar contexts globally, ultimately contributing to the global effort to reduce repeat adolescent pregnancy, improve mental health, and support the next generation of healthy, empowered mothers.

Important Administrative Note:

This study was originally registered under the administrative affiliation of Ross University School of Medicine (RUSM). While the study concept originated and was developed by the Sponsor-Investigator, the original IRB submission to RUSM experienced delays due to institutional backlog and administrative constraints. As of October 4, 2025, no participants have been enrolled under RUSM IRB oversight, and no data has been collected.

Following consultation with the Caribbean Public Health Agency Ethics Review Committee (CANREC), the Sponsor-Investigator was advised that ethical review and approval should be obtained through a local Institutional Review Board in Barbados. The study will not proceed until local IRB approval has been secured.

The Organization's Unique Protocol ID "RUSM20240405-CANREC20250903" reflects the administrative history of the project, including initial registration under RUSM on April 5, 2024, and subsequent guidance provided by CANREC beginning September 3, 2025. This identifier is maintained for administrative continuity only.

ELIGIBILITY:
Inclusion Criteria:

* Young mothers aged 10 to 25 years residing in Barbados
* Experienced adolescent pregnancy between ages 10 and 19 years
* Living in low-income households with annual income BDS $20,000 (~USD 10,000) or below
* Screen positive for depressed mood symptoms using the Patient Health Questionnaire-2 (PHQ-2), indicating feeling "little interest or pleasure in doing things" and/or feeling "down, depressed, or hopeless" over the past 2 weeks
* Able to provide informed consent or assent (with parental consent if under legal age)
* Willing to complete study questionnaires and attend scheduled visits

Exclusion Criteria:

* History of heart disease, head trauma, hypertension, diabetes, psychiatric, or neurological conditions
* Severe cognitive or medical conditions preventing participation
* Enrollment in conflicting interventional studies
* Insufficient proficiency in study languages without access to interpretation (if applicable)

Ages: 10 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Eligibility is based on biological sex, not gender identity.
Enrollment: 50 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure (mmHg) | At baseline and each site visit (e.g., bi-monthly for 6 months)
  Systolic blood pressure will be measured using a calibrated sphygmomanometer or automated device after participants have been seated and rested for 5 minutes.
Diastolic Blood Pressure (mmHg) | At baseline and each site visit (e.g., bi-monthly for 6 months)
  Diastolic blood pressure will be measured using the same method and protocol as systolic pressure.
  Unit of Measure: mmHg
Heart Rate (bpm) | At baseline and each site visit (e.g., bi-monthly for 6 months)
  Heart rate will be measured in beats per minute using standard clinical methods.
  Units: Beats per minute (bpm)
Respiration Rate (breaths per minute) | At baseline and each site visit (e.g., bi-monthly for 6 months)
  Respiration rate will be measured as the number of breaths per minute.
Glucose Level (mg/dL) | At baseline and each site visit (e.g., bi-monthly for 6 months)
  Blood glucose level will be measured via fingerstick or venous blood sample. Units: Milligrams per deciliter (mg/dL).
Body Temperature (°C) | At baseline and each site visit (e.g., bi-monthly for 6 months)
  Body temperature will be measured using a clinical thermometer (oral or tympanic) in degrees Celsius.
  Units: Degrees Celsius (°C)
Overall Health related to Mood-related symptoms Assessed by Patient Health Questionnaire-9 (PHQ-9) [Score Range: 0-27, Higher Scores Indicate Worse Outcome] | At baseline, each site visit (e.g., bi-monthly for 6 months), and 6 months post-intervention
  Overall health related to mood-related symptoms will be assessed using the Patient Health Questionnaire-9 (PHQ-9), a 9-item self-report scale assessing frequency of depressive-like symptoms over the past two weeks. Each item is scored from 0 (Not at all) to 3 (Nearly every day), producing a total score range of 0 to 27. Higher scores indicate more severe depression.
  Unit of Measure: PHQ-9 total score (0-27)
State Anxiety - State-Trait Anxiety Inventory (STAI or STAI-CH) | At baseline, week 24, and 6 months post-intervention
  STAI (or STAI-CH for adolescents) is a 20-item scale assessing anxiety symptoms.
  Min Score: 20. Max Score: 80. Higher scores indicate greater anxiety.
Depressive Symptoms in Adolescents - Center for Epidemiologic Studies Depression Scale (CES-D) | At baseline, week 24, and 6 months post-intervention
  A 20-item validated scale used widely in adolescent and pregnant populations.Min Score: 0. Max Score: 60. Higher scores indicate more depressive symptoms.
Parenting Stress - Parenting Stress Index (PSI) Short Form | At baseline, week 24, and 6 months post-intervention
  Measures perceived stress related to parenting using the PSI-SF, a 36-item validated tool.
  Min Score: 36. Max Score: 180. Higher scores indicate higher levels of stress.
Parenting Attitudes and Beliefs - Adult-Adolescent Parenting Inventory (AAPI-2) | Baseline and through study completion, an average of 1 year
  he AAPI-2 measures parenting beliefs and risk of abusive or harmful parenting practices.
  Min Score: 40. Max Score: 200. Higher scores indicate more appropriate/positive parenting attitudes.
Postpartum Social Support - Custom Self-Report Composite | Baseline, Week 12, and Week 24
  A composite measure including self-report variables on school status, repeat pregnancy, abuse history, substance use, and access to care.
  Unit of Measure: Categorical and descriptive data (each item analyzed separately)
Height (cm) | Baseline, Week 24
  Height will be measured using a stadiometer. Units: centimeters (cm)
Weight (lbs) | At baseline and each site visit (e.g., bimonthly for 6 months)
  Weight will be measured using a calibrated scale. Units: pounds (lbs)

SECONDARY OUTCOMES:
Changes in healthcare utilization | Through study completion, an average of 12 months
  Frequency of clinic visits, emergency room visits, and use of preventive health services over the study period.
  Unit of Measure: Number of visits per participant.
Child Developmental Outcomes - Ages and Stages Questionnaire (ASQ) | At 6 months and 12 months postpartum
  Physical, emotional, and cognitive development milestones assessed via the Ages and Stages Questionnaire.
  Min Score: 0.
  Max Score: Varies by domain and age.
  Higher scores indicate more age-appropriate development.
Child Growth - Weight (kg) | At 6 months and 12 months postpartum
  Weight of the child measured using standard pediatric scales. Unit of Measure: Kilograms
Child Growth - Height (cm) | At 6 months and 12 months postpartum
  Height/length of the child measured using standard equipment. Unit of Measure: Centimeters
Incidence of repeat pregnancy within study period | Up to 12 months postpartum
  Number of participants experiencing repeat pregnancies during the study timeframe.
Mental health service utilization | through study completion, an average of 1 year
  Frequency of use of mental health services, including therapy, counseling, or psychiatric care. Unit of Measure: Number of visits per participant.
Changes in Knowledge and Attitudes Toward Contraception and Sexual Health - THRIVE KASH-Q | through study completion, an average of 1 year
  A THRIVE-developed questionnaire measuring knowledge of and attitudes toward contraception and sexual health. Min Score: 0.
  Max Score: 100.
  Higher scores indicate better knowledge and more positive attitudes.
Satisfaction with Communication with healthcare providers in Integrated Care Model | Week 24
  Participant satisfaction with communication with healthcare providers will be assessed using a standardized 7-point Likert scale survey ranging from 1 (Completely Dissatisfactory), 2 (Moderately Dissatisfactory), 3 (Slightly Dissatisfactory), 4 (Neutral), 5 (Slightly Satisfactory), 6 (Moderately Satisfactory), to 7 (Completely Satisfactory) in a survey. Higher scores represent higher overall satisfaction.
Satisfaction with Access to Care in Integrated Care Model | Week 24
  Participant satisfaction with access to care will be assessed using a standardized 7-point Likert scale survey ranging from 1 (Completely Dissatisfactory), 2 (Moderately Dissatisfactory), 3 (Slightly Dissatisfactory), 4 (Neutral), 5 (Slightly Satisfactory), 6 (Moderately Satisfactory), to 7 (Completely Satisfactory) in a survey. Higher scores indicate greater satisfaction.
Satisfaction with Care Coordination in Integrated Care Model | Week 24
  Participants will rate their satisfaction with the coordination of the modules provided using a standardized 7-point Likert scale survey ranging from 1 (Completely Dissatisfactory), 2 (Moderately Dissatisfactory), 3 (Slightly Dissatisfactory), 4 (Neutral), 5 (Slightly Satisfactory), 6 (Moderately Satisfactory), to 7 (Completely Satisfactory) in a survey. Higher scores indicate greater satisfaction.
Satisfaction with Responsiveness to needs in Integrated Care Model | Week 24
  Participant satisfaction with responsiveness to participant's needs will be assessed using a standardized 7-point Likert scale survey ranging from 1 (Completely Dissatisfactory), 2 (Moderately Dissatisfactory), 3 (Slightly Dissatisfactory), 4 (Neutral), 5 (Slightly Satisfactory), 6 (Moderately Satisfactory), to 7 (Completely Satisfactory) in a survey. Higher scores represent higher overall satisfaction.
Overall Satisfaction with Integrated Care Model | Week 24
  Overall satisfaction with the integrated care model will be assessed using a standardized 7-point Likert scale survey ranging from 1 (Completely Dissatisfactory), 2 (Moderately Dissatisfactory), 3 (Slightly Dissatisfactory), 4 (Neutral), 5 (Slightly Satisfactory), 6 (Moderately Satisfactory), to 7 (Completely Satisfactory) in a survey. Higher scores represent higher overall satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Hada Fongha Ieong, PhD, Principal Investigator
Locations (1):
- Rotary Club of Barbados, Bridgetown, Barbados

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the sensitive nature of the study population and data. This trial involves adolescents and young adults, many of whom are minors, and collects sensitive information on reproductive health, mental health, and social risk factors. Ensuring participant privacy and confidentiality is a top ethical priority. At this time, there is no IRB-approved protocol or infrastructure in place for secure IPD sharing.

REFERENCES:
- [Result] Ieong HF, Cobbin M, Tlachi P, Chidsey C, Flaks R, Ross A. Barriers to randomized trials of integrated care for adolescent mothers in the Caribbean: lessons from the THRIVE trial and the Project Amai in Barbados. Trials. 2025 Dec 17;27(1):65. doi: 10.1186/s13063-025-09359-8. PMID 41408317
- See also: Barriers to randomized trials of integrated care for adolescent mothers in the Caribbean: lessons from the THRIVE trial and the Project Amai in Barbados — https://doi.org/10.1186/s13063-025-09359-8